CLINICAL TRIAL: NCT05833646
Title: Comparison of the Effects of ShotBlocker, Virtual Reality Glasses and Cold Application on Pain and Patient Satisfaction in Subcutaneous Heparin Injection Application in Adult Patients
Brief Title: Comparison of the Effects of ShotBlocker, Virtual Reality Glasses and Cold Application in Subcutaneous Heparin Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ebru Erek Kazan, Assoc.Prof., Ankara Yildirim Beyazıt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1790
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Subcutaneous Injection
Keywords: Subcutaneous injection; Pain; Satisfaction; Virtual reality; ShotBlocker; Cold application; Nursing
MeSH Terms: conditions — Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Self-controlled, quasi-experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ShotBlocker Group (Experimental): In control application, subcutaneous (SC) LMWH injection will be applied in patient's left abdomen with standard method on Post-op 0th day by the researcher. Intervention with ShotBlocker will be performed on the right abdomen site on post-op 1st day by the researcher. During subcutaneous LMWH injection with ShotBlocker, suitable injection site in right abdomen will be grasped by applying medium-weight pressure as ShotBlocker's obtuse touching points would touch the skin. In order to avoid ecchymosis and hematoma, it will be applied slowly for 10 seconds by entering from the middle point of ShotBlocker with a 90° angle. When injection is over, ShotBlocker will be removed 10 seconds will be waited. Removing the needle, the entry point will be applied light pressure with dry cotton for 10 seconds without any massage. Patients' level of pain and satisfaction will be assessed by a nurse working in the clinic with visual analog scale (VAS) within 1 minute after injection.
  Interventions: Device: Group 1
- Virtual Reality Glasses (VRG) Group (Experimental): Standard LMWH application will be performed on the left side for control on Post-op 0th day by the researcher.
  Intervention with VRG will be performed on the right abdomen site on post-op 1st day. The researcher will show the patient a video 5 minutes before the injection providing them with virtual reality glasses, which will continue till the end of the operation, after which the glasses will be removed. Patients' level of pain and satisfaction will be assessed by a nurse working in the clinic with visual analog scale (VAS) within 1 minute after injection.
  Interventions: Device: Group 2
- Cold Application Group (Experimental): Standard heparin application will be performed on left side for control on post-op 0th day by the researcher. Intervention with cold application will be performed on the right abdomen site on post-op 1st day. Prior to the intervention, cold silica gel pack which stayed in the freezer for at least 2 hours will be placed on patient's injection site by wrapping up with towel and will be applied on the site for 5 minutes. After 5 minutes, the cold gel pack will be removed from the site and subcutaneous LMWH injection will be applied by the researcher. Following the removal of the injector, cold application will continue for another 2 minutes. Patients' level of pain and satisfaction will be assessed by a nurse working in the clinic with visual analog scale (VAS) after injection.
  Interventions: Device: Group 3

INTERVENTIONS:
Device: Group 1 — In each group, patients will be applied both standard subcutaneous heparin injection and with ShotBlocker.
  Other Names: ShotBlocker
  Arms: ShotBlocker Group
Device: Group 2 — In each group, patients will be applied both standard subcutaneous heparin injection and with virtual reality glasses.
  Other Names: Virtual Reality Glasses (VRG)
  Arms: Virtual Reality Glasses (VRG) Group
Device: Group 3 — In each group, patients will be applied both standard subcutaneous heparin injection and with cold application.
  Other Names: Cold Application
  Arms: Cold Application Group

SUMMARY:
This study aims to compare the effects of ShotBlocker, virtual reality glasses and cold application on pain and patient satisfaction in patients who were applied subcutaneous low molecular weight heparin (LMWH) injection in adult patients.

DETAILED DESCRIPTION:
The research being carried out in Ankara City Hospital Clinic of Orthopedics. The research sample is expected to consist of 150 adult patients, who will be randomly divided into three groups. First group will be applied ShotBlocker (n=50); second group will be applied Virtual Reality Glasses (n=50) and third group will be applied subcutaneous LMWH via cold application (n=50). So as to assess the effect of the injection, it will be applied on patients' left side within abdomen site via standard method (control) while the same will be done on patients' right side according to method of intervention (intervention). Therefore, each patient will form both intervention and control groups. Prior to subcutaneous LMWH injection, "Descriptive Characteristics Form", which includes participants' socio-demographic attributes (gender, marital status, age, level of education, etc.), will be filled out by the researcher by means of face-to-face interview. Following the injection, in order to evaluate patients' pain, "Visual Analog Scale for Pain" will be filled while "Visual Analog Scale for Satisfaction" will be used in order to identify patients' satisfaction with the application. It is expected that compared to standard injection, ShotBlocker, virtual reality glasses and cold application will reveal more positive results on pain and patient satisfaction during subcutaneous LMWH injection in adult patients. Besides, the method that has the more effect will be determined by comparing different methods. It is thought the data collected by the research will contribute to literature.

ELIGIBILITY:
Inclusion Criteria:

* Open to communication
* 18 or over years of age
* Received 1x0,4 ml enoksaparin sodium treatment
* Experienced no complications during or after operation
* Normal values of thrombocyte (150.000-300.000), aPTT (25-35 sec) and INR (0.8-1.2) (Thrombocyte, INR and aPTT tests will be assessed in accordance with reference values of the kits that the hospital uses.)
* No infection, scar tissue or incision in abdomen site
* Received no parenteral treatment other than this site
* Not diagnosed with any sort of coagulation disorder
* No visual impairment to be able to wear VR glasses
* No allergy to cold
* No mental or neurological disability
* No audio-visual impairment disability to be able to watch the video
* Turkish speaking and comprehending
* Non-pregnant
* No hematological or allergic disease
* Willing to be hospitalized for 2 days
* Volunteer to participate in the research will constitute the research sample.

Exclusion Criteria:

During data collection, those who;

* Renounce from participating in the research
* Remove virtual reality glasses during or after operation
* Fail to hold the cold pack for necessary period of time
* Show signs of cold allergy during operation
* Change institutions or were discharged early during research
* Change dose of drugs within drug system
* Develop drawbacks in the abdomen site will be excluded from the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Pain assessed by the VAS (Visual Analog Scale) | 4 month
  In this research, in order to assess patients' level of injection pain, Visual Analog Scale (VAS) will be used. It is a 10 cm scale, on each side of which there is "no pain" and "worst pain". In using VAS, the patient is informed that they are free to choose a spot between two endpoints and the destination from the start of "no pain" and the spot the patient chooses is measured and recorded as cm./ mm. In this assessment, mean pain scores ranging among 1-10 are given. Thus, while "0" refers to no pain, 1-4 VAS values refer to dull pain; 5-6 to moderate pain; 7-10 refer to worst pain. Results will be compared both within group and among all groups at the end of the research.
Satisfaction assessed by the VAS (Visual Analog Scale) | 4 month
  VAS is also used to measure components other than pain. VAS-Patient Satisfaction is a 10 cm scale, on each side of which there is "Dissatisfied" and "Very Satisfied". After injection, the patient is expect to detect their level of satisfaction by synthesizing affecting factors related to the process and mark the level of satisfaction on a line with a cross (X). High scores obtained from the scale refer to high levels of patient satisfaction. Results will be compared both within group and among all groups at the end of the research.

CONTACTS AND LOCATIONS:
Overall Officials: Hafize Güllü, MsN, Principal Investigator — Ankara Yildirim Beyazit University , Faculty of Health Sciences, Department of Nursing
Locations (1):
- Ankara Yildirim Beyazit University Faculty of Health Sciences, Department of Nursing, Ankara, Çubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No